CLINICAL TRIAL: NCT07013214
Title: Rehabilitation Program to Improve Balance in Patients With Parkinson's Disease: Dual-Task Exercise - A Randomized Controlled Clinical Trial
Brief Title: Rehabilitation With Dual-task Exercises to Improve Balance in Patients With Parkinson's Disease
Acronym: DUAL-PD-RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: G. d'Annunzio University (Other)
Responsible Party: Principal Investigator, Teresa Paolucci, Professor, MD, PhD, Physical Medicine and Rehabilitation Physician, G. d'Annunzio University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 180426/25; 237 (Other: Università degli Studi "G. d'Annunzio" Chieti - DSMOB)
Record Dates: First submitted 2025-06-02; First posted 2025-06-10 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Parkinson Disease (PD), Postural Balance
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dual-Task Exercise Program (Experimental): This arm consists of participants assigned to receive a structured rehabilitative pathway based on dual-task exercises. This program integrates motor and cognitive tasks simultaneously, and is designed to improve balance, reduce fall risk, and enhance autonomy and quality of life in Parkinson's patients. Participants in this group will complete a total of 20 sessions, administered 2-3 times per week for a duration of two months, with each session lasting 45 minutes.
  Interventions: Behavioral: Dual-Task Exercise
- Standard Rehabilitation Program (Active Comparator): This arm consists of participants assigned to receive a standard rehabilitation program. This intervention focuses on traditional motor rehabilitation techniques and serves as the active control group for comparison with the dual-task intervention. Participants in this group will complete a total of 20 sessions, administered 2-3 times per week for a duration of two months, with each session lasting 45 minutes.
  Interventions: Behavioral: Standard Rehabilitation

INTERVENTIONS:
Behavioral: Dual-Task Exercise — This intervention consists of exercises that integrate motor tasks (e.g., balance training, walking) with concurrent cognitive tasks (e.g., counting, verbal fluency, decision-making tasks). The progression of exercises will be tailored to the individual's abilities, gradually increasing the difficulty of both the motor and cognitive components.
  Arms: Dual-Task Exercise Program
Behavioral: Standard Rehabilitation — This intervention consists of conventional exercises aimed at improving balance, gait, posture, and flexibility, without the integration of simultaneous cognitive tasks. The program will focus on established physical therapy techniques for Parkinson's disease.
  Arms: Standard Rehabilitation Program

SUMMARY:
The goal of this clinical trial is to learn if a rehabilitative pathway based on dual-task exercise improves balance in patients with Parkinson's disease, compared to a traditional rehabilitation program. It will also investigate the reduction of fall risk, and improvement in autonomy and quality of life.

The main questions it aims to answer are:

* Does dual-task exercise improve balance more effectively than traditional rehabilitation in Parkinson's patients?
* Does dual-task exercise reduce the risk of falls?
* Does dual-task exercise improve patient autonomy in daily activities?
* Does dual-task exercise enhance the overall quality of life for Parkinson's patients? Researchers will compare a dual-task exercise program to a standard rehabilitation program. Both groups will receive 20 sessions, 2-3 times a week for two months, each lasting 45 minutes. The study will be double-blinded, meaning neither participants nor researchers involved in treatment administration and data collection will know group assignments. Randomization will be done using dedicated software to ensure unbiased group distribution.

Participants will:

* Have a confirmed diagnosis of Parkinson's disease (Movement Disorder Society criteria).
* Be in an early to moderate stage of the disease (Hoehn and Yahr score < 3).
* Be over 30 years old.
* Be able to provide informed consent.
* Have a stable medication regimen for at least three months.

Exclusions include:

* Hoehn and Yahr score ≥3.
* Severe cognitive or psychiatric disorders (e.g., dementia).
* Use of interfering medications or treatments.
* Participation in other clinical trials.
* Pregnancy or breastfeeding.
* Need for medication changes during rehabilitation. Evaluations will be conducted at baseline (T=0), after rehabilitation (T=1), and at a two-month follow-up (T=2). Assessments will include the Tinetti Balance and Gait scales, Timed Up and Go (TUG) test, VAS pain scale, TAMPA Scale for Kinesiophobia, Global Perceived Effect (GPE), Barthel Index, EuroQoL-5D-5L, and ABC Scale. UPDRS, Hoehn and Yahr scale, and MOCA Scale will be administered only at baseline (T=0).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Parkinson's Disease (Movement Disorder Society criteria).
* Early to moderate stage of the disease (Hoehn and Yahr score < 3).
* Age over 30 years.
* Ability to provide informed consent.
* Stable pharmacological therapy for at least 3 months.

Exclusion Criteria:

* Hoehn and Yahr score ≥ 3.
* Severe cognitive or psychiatric disorders (e.g., dementia).
* Use of interfering medications or treatments.
* Participation in another clinical trial.
* Pregnancy or breastfeeding.
* Need for changes in pharmacological therapy during the rehabilitation period.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2025-07-07 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
UPDRS (Unified Parkinson's Disease Rating Scale) | Baseline
  It is a widely used scale to assess the severity of symptoms in patients with Parkinson's disease. It consists of four sections: non-motor and mental aspects, motor aspects, motor complications, and treatment. It evaluates aspects such as tremor, rigidity, bradykinesia, balance, and daily activities.
Hoehn and Yahr scale | Baseline
  It is a staging scale that classifies the severity of Parkinson's disease into five stages, from mild (stage 1) to severe (stage 5), based on the presence of motor symptoms and functional impairment.
MOCA Scale (Montreal Cognitive Assessment) | Baseline
  The MoCA is a screening tool used to assess cognitive functions. It is designed to detect mild and moderate cognitive impairments, such as those associated with dementia or other neurological conditions. The scale covers various cognitive domains, including attention, concentration, memory, language, visuospatial abilities, abstraction, calculation, and orientation. The maximum score is 30 points, and a score below 26 may indicate the presence of cognitive impairment.
Tinetti Balance and Gait scales | -At study enrollment (Baseline) -Immediately after completion of the 2-month rehabilitation program -At 2-month follow-up after rehabilitation program completion
  Two distinct but related scales:
  * Tinetti Balance Scale: assesses fall risk through various balance tests.
  * Tinetti Gait Scale: evaluates gait and the related risk of falling. Both scales are used to identify individuals at risk of falling and to monitor the effectiveness of interventions.
TUG (Timed Up and Go test) | -At study enrollment (Baseline) -Immediately after completion of the 2-month rehabilitation program -At 2-month follow-up after rehabilitation program completion
  It is a simple test that measures the time a person takes to stand up from a chair, walk three meters, turn around, return, and sit down. It is used to assess balance and fall risk.

SECONDARY OUTCOMES:
Visual Analogue Scale for pain (VAS) | -At study enrollment (Baseline) -Immediately after completion of the 2-month rehabilitation program -At 2-month follow-up after rehabilitation program completion
  It is a subjective scale that allows patients to rate their level of pain on a 10 cm line, where 0 indicates no pain and 10 indicates the worst imaginable pain.
TAMPA Scale (Tampa Scale for Kinesiophobia) | -At study enrollment (Baseline) -Immediately after completion of the 2-month rehabilitation program -At 2-month follow-up after rehabilitation program completion
  It assesses the fear of movement or reactivation due to pain or risk of injury. It consists of questions that measure the fear of moving and becoming active again.
Global Perceived Effect (GPE) | -At study enrollment (Baseline) -Immediately after completion of the 2-month rehabilitation program -At 2-month follow-up after rehabilitation program completion
  It is a subjective scale used to assess a patient's overall perception of improvement or worsening after an intervention or treatment. A 7-point scale is typically used, where the patient indicates whether they feel much improved, improved, unchanged, worsened, or much worsened. It is a simple and quick tool to obtain a global assessment of the perceived effectiveness of the treatment.
Barthel Index | -At study enrollment (Baseline) -Immediately after completion of the 2-month rehabilitation program -At 2-month follow-up after rehabilitation program completion
  It is a scale used to assess the level of independence in activities of daily living (ADLs). It includes 10 items covering activities such as eating, dressing, personal hygiene, mobility, using the toilet, continence, and walking or moving around. Each activity is scored, contributing to a total maximum score of 100, where a higher score indicates greater independence.
EuroQoL-5D-5L (EuroQoLD5L) | -At study enrollment (Baseline) -Immediately after completion of the 2-month rehabilitation program -At 2-month follow-up after rehabilitation program completion
  It is a tool used to assess health-related quality of life. It includes five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has five levels of severity, ranging from no problems to extreme problems. In addition, it includes a visual analogue scale (VAS) where the patient rates their overall health on a scale from 0 to 100. It is widely used in clinical research and public health assessments.
ABC Scale (Activities-specific Balance Confidence Scale) | -At study enrollment (Baseline) -Immediately after completion of the 2-month rehabilitation program -At 2-month follow-up after rehabilitation program completion
  It measures the patient's confidence in their ability to maintain balance during various daily activities. It consists of 16 items, each rated on a scale from 0% (no confidence) to 100% (complete confidence). It is particularly useful for assessing fall risk and the effectiveness of rehabilitation interventions aimed at improving balance and safety in daily activities.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Paolo Sesto - Centro Adriatico, Pescara, PE, Italy

IPD SHARING:
Plan to Share IPD: Yes